CLINICAL TRIAL: NCT05114096
Title: Single Dose of Antenatal Corticosteroids (SNACS) Randomized Controlled Trial for Pregnancies at Risk of Preterm Delivery: To Keep Babies and Children Safe
Brief Title: Single Dose of Antenatal Corticosteroids for Pregnancies at Risk of Preterm Delivery (SNACS)
Acronym: SNACS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Sunnybrook Research Institute (Other); Women's and Children's Hospital, Australia (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); Medical Research Future Fund (Other); University of Adelaide (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 3764
Record Dates: First submitted 2021-10-12; First posted 2021-11-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Preterm Birth; Premature Birth; Complication of Prematurity; Obstetric Labor, Premature; Pregnancy Complications
Keywords: Premature birth; Preterm birth; Obstetric labour; Betamethasone; Betamethasone Valerate; Betamethasone-17,21-dipropionate; Betamethasone benzoate; Betamethasone sodium phosphate; Anti-Inflammatory Agents; Glucocorticoids; Hormones; Hormones, Hormone Substitutes and Hormone Antagonists; Physiological Effect of Drugs; Anti-Asthmatic Agents; Respiratory System Agents
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Pregnancy Complications | interventions — Betamethasone

STUDY DESIGN:
Intervention Model Description: Multicentre, blinded, pragmatic, 2 arm non-inferiority RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-Dose Celestone (Experimental): Having already received the first dose of Celestone as part of eligibility criteria, participants randomized to the experimental "Single-Dose" arm will receive a similar appearing placebo injection.
  Interventions: Drug: Celestone + placebo
- Double-Dose Celestone (Active Comparator): Having already received the first dose of Celestone as part of eligibility criteria, participants randomized to the "Double-Dose" arm will receive the standard 2nd dose of Celestone injected intramuscularly (i.e. they will receive the standard double-dose regimen).
  Interventions: Drug: Celestone + Celestone

INTERVENTIONS:
Drug: Celestone + placebo — After the first intramuscular injection of Celestone, participants randomized to the "Placebo Comparator" group will receive 1 intramuscular injection of placebo.
  Arms: Single-Dose Celestone
Drug: Celestone + Celestone — After the first intramuscular injection of Celestone, participants randomized to the "Active Comparator" group will receive 1 intramuscular injection of Celestone.
  Arms: Double-Dose Celestone

SUMMARY:
Antenatal corticosteroids (ACS) reduce the risks of neonatal death and morbidities in preterm infants, such as respiratory distress syndrome.

The standard of care for pregnant people at risk of preterm birth includes 2 doses of Celestone (for a total of 24 mg in Canada, or 22.8 mg in Australia) to accelerate fetal lung maturity.

The investigators plan to conduct a randomized controlled trial to determine whether half the usual dose (12 mg in Canada, or 11.4 mg in Australia) of Celestone is non-inferior to the standard double doses.

DETAILED DESCRIPTION:
Preterm infants are at risk of mortality and morbidity. Antenatal corticosteroids (ACS) reduce the risks of neonatal death and morbidities, such as respiratory distress syndrome.

The standard of care for pregnant people at risk of preterm birth includes 2 doses of Celestone to accelerate fetal lung maturity (total 24 mg in Canada, 22.8 mg in Australia). There are no published clinical trial data on the benefits or risks of a single dose of antenatal corticosteroid vs. standard double doses (Ninan et al JOGC 2020).

Pregnant people at 22 weeks and 0 days to < 34 weeks and 6 days' gestation at risk of preterm birth with a singleton or twin gestation who have received the first dose of Celestone and consented to the trial will be randomized to receive approximately 24 hours later either an experimental placebo injection (of normal saline) or the standard double dose of Celestone to determine whether the intervention is non-inferior for the primary outcome of a composite of perinatal mortality or substantial morbidity.

Please note: Based on Health Canada's' guidance the study phase is 'Other: Off-Label use'. However, on the clincaltrial.gov record, 'Phase 4' is selected as this is the most relevant phase and there is no option to select 'Other'.

Please note: McMaster University, Canada is the Canadian Regulatory Sponsor and Overall Sponsor, and the University of Adelaide Australia is the Australian Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant people, aged 18 to 55 years old, at risk of preterm birth with a singleton or twins between 22 weeks and 0 days and <34 weeks and 6 days gestation who have received only a single dose of Celestone within 24 hours
2. Capable of giving informed, written consent.

Exclusion Criteria:

1. Contraindication to corticosteroids
2. Systemic corticosteroids for medical conditions during the pregnancy (e.g. lupus, severe asthma, Covid, etc).
3. Previous participation in this trial (in a previous pregnancy)
4. Known severe/life-threatening fetal or pregnant patient condition (e.g. fetal congenital/chromosomal abnormality)
5. Demise of one or more fetuses after 14 weeks and 0 days

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3254 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Perinatal Mortality or Substantial Neonatal Morbidity | approximately 1 month
  Fetal death post-randomization or in hospital neonatal death OR => 1 of respiratory morbidity (requiring surfactant <=48 hrs of life), severe intraventricular hemorrhage (distending/beyond the ventricles, i.e. Grade 3 or 4), or severe bowel problem (necrotizing enterocolitis, Stage 2 or 3)

SECONDARY OUTCOMES:
Death or neurosensory/developmental impairment at 24 months | approximately 24 months
  Death or neurosensory/developmental impairment at 24 months (+/- 6 months; accounting for gestation at birth), mood (anxiety/depression), behavior (aggression), etc as assessed by:
  1. Ages and Stages Questionnaire-3 (ASQ)
  2. Child Behavior Checklist: 4 subscales
  3. Physician diagnosis of cerebral palsy (parent report).

OTHER OUTCOMES:
Number of babies who received intubation and duration of invasive mechanical ventilation | approximately up to first 6 months of life
  Number of babies who received intubation and duration of invasive mechanical ventilation
Number of babies who received, and duration of, supplemental oxygen (after resuscitation) and other ventilatory support | approximately up to first 6 months of life
  Number of babies who received, and duration of, supplemental oxygen (after resuscitation) and other ventilatory support
Number of babies with respiratory distress after the initial resuscitation/stabilization and main cause | approximately 1 month
  Number of babies with respiratory distress after the initial resuscitation/stabilization and main cause (such as respiratory distress syndrome, pneumothorax/pneumomediastinum, pneumonia, transient tachypnea of the newborn, meconium aspiration syndrome, persistent pulmonary hypertension of the newborn)
Number of babies with Respiratory distress after the initial resuscitation/stabilization and main cause | approximately at birth
  Respiratory distress after the initial resuscitation/stabilization and main cause (such as respiratory distress syndrome, pneumothorax/pneumomediastinum, pneumonia, transient tachypnea of the newborn, meconium aspiration syndrome, persistent pulmonary hypertension of the newborn),
Number of babies with hypoglycemia | 48 hours
  Number of babies with hypoglycemia (low plasma glucose < 2.6 mmol/L between 30 minutes and 48 hours of life)
Number of babies with neonatal sepsis | 7 days
  Number of babies with neonatal sepsis within 7 days of birth, defined as a positive (bacterial, viral or fungal): blood culture or cerebrospinal fluid culture (or gram stain) or urine culture by sterile collection.
Number of babies with severe retinopathy of prematurity needing treatment | approximately first few months of life
  Number of babies with severe retinopathy of prematurity defined as requiring vascular endothelial growth factor (VEGF) or laser or cryotherapy per the local guidelines
Number of babies with patent ductus arteriosus (PDA) needing a closure procedure (surgery or device) | up to 12 weeks after birth
  Number of babies with patent ductus arteriosus (PDA) needing a closure procedure (surgery or device)
Anthropometry at birth and at 24 months corrected age | at birth and at 24 months corrected age
  Weight (in grams), length (in centimeters), and head circumference (in centimeters) for birth week as ACS can impact growth
Number of babies with severe late brain injury | up to 20 weeks postnatal
  Periventricular leukomalacia [PVL], i.e. cystic changes in white matter or porencephalic cysts or white matter changes diagnosed by ultrasound or MRI.
Number of babies with chronic lung disease | approximately up to first 6 months of life
  Late respiratory morbidity, bronchopulmonary dysplasia (BPD), defined as requiring respiratory support or supplemental oxygen > 36 completed weeks' corrected gestation.
Apgar score and cord blood pH | approximately at birth
  Apgar score (at 1 and 5 min) and lowest cord blood pH, regardless of whether arterial or venous.
Length of stay in special care or an intensive care setting | approximately up to first 6 months of life
  Length of stay in an intensive care setting such as the neonatal intensive care unit (NICU).
Use of postnatal corticosteroids | up to 20 weeks postnatal
  Use of systemic (intravenous or oral) postnatal corticosteroids and type (e.g. hydrocortisone, dexamethasone).
Number of babies with longterm health care outcomes | approximately 5 -10 years
  Number of babies with reported longterm health care outcomes after initial hospital, such as hospitalizations, and other health care use.
Number of babies with longterm education outcomes | approximately 5 -10 years
  Number of babies with reported longterm education or non-health data outcomes, collected through database linkage where possible.
Number of participants with fetal death post-randomization or in hospital neonatal death OR => 1 of respiratory morbidity, severe intraventricular hemorrhage , or severe bowel problem | approximately 1 month
  Fetal death post-randomization or in hospital neonatal death OR => 1 of respiratory morbidity (requiring surfactant <=48 hrs of life), severe intraventricular hemorrhage (distending/beyond the ventricles, i.e. Grade 3 or 4), or severe bowel problem (necrotizing enterocolitis, Stage 2 or 3)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D McDonald, MD,MSc,FRCSC, Principal Investigator — McMaster University; Kellie Murphy, MD,MSc,FRCSC, Principal Investigator — University of Toronto
Locations (25):
- Canada (25):
  - University of Calgary, Cumming School of Medicine, Calgary, Alberta
  - Alberta Health Services; University of Alberta, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Fraser Health, University of British Columbia; Jim Pattison Outpatient Care and Surgery Centre, Surrey, British Columbia
  - University of British Columbia; BC Women's Hospital, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - University of Manitoba, Health Sciences Centre, Winnipeg, Manitoba
  - University of Manitoba; St. Boniface General Hospital, Winnipeg, Manitoba
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - The Moncton Hospital, Horizon Health Network, Moncton, New Brunswick
  - Memorial University, Eastern Health, St. John's, Newfoundland and Labrador
  - Dalhousie University; Izaak Walton Killam Health, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston General Hospital Health Sciences Centre, Kingston, Ontario
  - Western University; London Health Sciences Centre, Victoria Hospital, London, Ontario
  - University of Ottawa; The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, CIUSSS de l'est de l'Ile de Montréal, Montreal, Quebec
  - McGill University, McGill University Health Center, Royal Victoria Hospital, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital; McGill University, Montreal, Quebec
  - The Centre Hospitalier Universitaire Sainte-Justine, Université de Montréal, Montreal, Quebec
  - Université Laval, Centre de recherche du CHU de Québec, Québec, Quebec
  - (CIUSSS de l'Estrie-CHUS); Université de Sherbrooke, Sherbrooke, Quebec
  - University of Saskatchewan, Regina General Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
An IPD is planned with trial leaders of another half dose Celestone study.

REFERENCES:
- [Background] Ninan K, Morfaw F, Murphy KE, Beyene J, McDonald SD. Neonatal and Maternal Outcomes of Lower Versus Standard Doses of Antenatal Corticosteroids for Women at Risk of Preterm Delivery: A Systematic Review of Randomized Controlled Trials. J Obstet Gynaecol Can. 2021 Jan;43(1):74-81. doi: 10.1016/j.jogc.2020.02.127. Epub 2020 Mar 26. PMID 32660867
- See also: Neonatal and Maternal Outcomes of Lower Versus Standard Doses of Antenatal Corticosteroids for Women at Risk of Preterm Delivery: A Systematic Review of Randomized Controlled Trials — https://doi.org/10.1016/j.jogc.2020.02.127